CLINICAL TRIAL: NCT03161054
Title: A Phase II Study of Metronomic Chemotherapy in Elderly Non-fit Patients (>65 Years) With Aggressive B-Cell Lymphomas
Brief Title: Metronomic Chemotherapy in Elderly Non-fit Patients With Aggressive B-Cell Lymphomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_DEVEC
Record Dates: First submitted 2017-05-18; First posted 2017-05-19 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Aggressive Non-Hodgkin Lymphoma
Keywords: Metronomic Chemotherapy; Elderly non-fit patients; Aggressive B-Cell lymphomas
MeSH Terms: interventions — Prednisone; Vinorelbine; Etoposide; Cyclophosphamide; Rituximab

STUDY DESIGN:
Intervention Model Description: phase II, multicentre, non-randomized study, single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One arm for all patient (Experimental): Induction phase:
  Eligible Pts will receive 6 cycles (every 28 days) of the DEVEC combination: DE: Prednisone, V: Vinorelbine, E: Etoposide, C: Cyclophosphamide and R:Rituximab ; R will be administered only in patients suitable for infusion treatment and relapsed after >6 months from last R-chemotherapy. Refractory patients who received at least 5 doses of R will not repeat it during the metronomic therapy.
  Super-frail patients will not receive etoposide during cycles 1 and 2.
  Maintenance Phase:
  Pts in CR, CRu and PR at the end of the induction phase, will continue treatment with maintenance therapy including Vinorelbine, Cyclophosphamide, and Prednisone oral combination to be repeated every 28 days for up to 6 cycles.
  Post Maintenance Phase:
  Pts in CR/CRu at the EOT may, at discretion of the local investigator, continue maintenance with only Vinorelbine and Prednisone for up to further 12 months, progression or inacceptable toxicity at the same doses of maintenance
  Interventions: Drug: Prednisone; Drug: Vinorelbine; Drug: Etoposide; Drug: Cyclophosphamide; Drug: Rituximab

INTERVENTIONS:
Drug: Prednisone — Induction Phase: Prednisone (Deltacortene) 25 mg /day will be orally administered from day 1 to day 28 only in cycle 1 From cycle 2 to 6 reduce to three times a week (after breakfast).
  Maintenance Phase: Prednisone 25 mg/day will be orally administered twice a week continuously (after breakfast).
  Post Maintenance Phase: Prednisone 25 mg/day will be orally administered twice a week continuously (after breakfast).
Drug: Vinorelbine — Induction Phase: Vinorelbine 30 mg/day will be orally administered three times a week, 3 weeks on and 1 week off (after breakfast).
  Maintenance Phase: Vinorelbine 30 mg/day will be orally administered three times a week, 3 weeks on and 1 week off (after breakfast).
  Post Maintenance Phase: vinorelbine 30 mg/day will be orally administered three times a week, 3 weeks on and 1 week off (after breakfast).
Drug: Etoposide — Induction Phase Etoposide: 50 mg/day will be orally administered from day 1 to day 14 (before lunch); Superfrail patients only from cycle 3, 50 mg/day, from day 1 to day 7
Drug: Cyclophosphamide — Induction Phase: Cyclophosphamide 50 mg/day will be orally administered from day 1 to day 21 (after dinner).
  Maintenance Phase: 50 mg/day will be orally administered from day 1 to day 14 (after dinner).
Drug: Rituximab — Induction Phase: Rituximab: 375 mg/m2 will be administered by IV infusion up to four infusions on days 8, 15, 22, 29, only in patients suitable for infusion treatment and relapsed after >6 months from last R-chemotherapy. Refractory patients who received at least 5 doses of Rituximab will not repeat it during the metronomic therapy.

SUMMARY:
This is a phase II study of metronomic chemotherapy in elderly non-fit patients (>65 years) with aggressive B-Cell lymphomas

DETAILED DESCRIPTION:
Patients eligible for the study will receive 6 courses (q 28 days) of the DEVEC combination, according to the following schedule:

* DE: Prednisone (Deltacortene) 25 mg /day will be orally administered from day 1 to day 28 only in cycle 1 From cycle 2 to 6 it is reduced to three times a week (after breakfast, MON, WED, FRI)
* V: Vinorelbine 30 mg/day will be orally administered three times a week, 3 week on and 1 week off (after breakfast, MON, WED, FRI).
* E: Etoposide 50 mg/day will be orally administered from day 1 to day 14 (before lunch).
* C: Cyclophosphamide 50 mg/day will be orally administered from day 1 to day 21 (after dinner).
* Rituximab: 375 mg/m2 will be administered by IV infusion up to four infusions on days 8, 15, 22, 29, only in patients suitable for infusion treatment and relapsed after >6 months from last R-chemotherapy. Refractory patients who had received at least 5 doses of Rituximab will not repeat it during the metronomic therapy.

Super-frail patients will not receive etoposide during cycles 1 and 2; etoposide will be included in the treatment schedule starting from cycle 3 at reduced dose (50 mg/day, from day 1 to day 7) only in patients who in cycles 1 and 2 didn't experience hematological toxicity >G2 and/or non-hematological toxicity >G1.

In Unfit and Frail patients with hemoglobin level at study entry <11 gr/dL, will start etoposide will be orally administered at reduced dose (50 mg/day from day 1 to day 7). If hemoglobin will raise to ≥11 gr/dL, at subsequent induction cycles etoposide will be administered at full dose (50 mg/day, from day 1 to day 14), As a preventive measure, to avoid perforation, patients with gastrointestinal visceral involvement will receive a pre-phase therapy with steroids (prednisolone 40mg/m2

) for 6-7 days before starting protocol treatment. Moreover, in these patients the four Rituximab doses will be administered in cycle 2.

Patients in CR, CRu, PR and SD after 2 cycles will continue with additional 4 courses.

At the end of the induction phase patients in CR, CRu and PR (and also in SD at discretion of local investigator) will continue treatment with maintenance therapy including Vinorelbine, Cyclophosphamide, and Prednisone oral combination to be repeated every 28 days for up to 6 cycles, according to the following schedule:

* Cyclophosphamide 50 mg/day will be orally administered from day 1 to day 14 (after dinner).
* Vinorelbine 30 mg/day will be orally administered three times a week, 3 week on and 1 week off (after breakfast, MON, WED, FRI).
* Prednisone 25 mg/day will be orally administered twice a week (after breakfast, MON, FRI).

Patients in CR/CRu at the EOT can continue with a post-maintenance phase at discretion of the local investigator up to 12 months, progression or inacceptable toxicity, according to following schedule:

* Vinorelbine 30 mg/day will be orally administered three times a week, 3 week on and 1 week off (after breakfast, MON, WED, FRI).
* Prednisone 25 mg/day will be orally administered twice a week (after breakfast, MON, FRI).

Patients with evidence of Progressive Disease (PD) at any point will stop treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of aggressive Non-Hodgkin Lymphomas (NHLs) including:

  * LBCL1
  * DLBCL;
  * Grade IIIb follicular lymphoma;
  * BL1;
  * B-Cell unclassifiable lymphomas with features intermediate between DLBCL and BL or between DLBCL and Hodgkin's lymphoma (HL)35;
  * High grade B-cell lymphomas1
* Age >65 years
* Unfit or frail patients (the latest defined, for the purpose of this study, as those who have a maximum of 1 frail factor) according to the multidimensional geriatric evaluation model of the elderly platform of the FIL, who relapsed/progressed after one or maximum two previous lines of treatment or
* "Super-frail" elderly patients at disease onset: eligible super-frail patients are defined, for the purpose of this study, as those who have a maximum of 2 frail factors, according to the CGA adopted in the elderly platform of the FIL, among those below listed:

  * ADL ≤ 4;
  * IADL ≤ 5;
  * Age ≥ 80 years;
  * 1 CIRS grade 3 or >8 CIRS grade 2.
* Ann Arbor stage I bulky to IV
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Life expectancy >1-2 months.
* Adequate renal function (creatinine ≤ 2 mg/dl, unless secondary to lymphoma).
* Adequate liver function (bilirubin ≤ 2 mg/dl, unless secondary to lymphoma).
* Absolute neutrophil count (ANC) ≥1500 cells/mmc and platelets ≥ 50,000 cells/mmc, haemoglobin ≥ 9 gr/dl, unless cytopenia is related to bone marrow involvement by lymphoma.
* Availability of adequate care by family members or other caregivers.
* Written informed consent signature.
* Male Subjects must agree to use a latex condom during sexual contact with females of childbearing potential while participating in the study and for at least 3 months following the end or the discontinuation from the study treatment even if he has undergone a successful vasectomy.

Exclusion Criteria:

* Patients who received more than two previous chemotherapy lines.
* Relapsed/refractory patients with fit profile.
* Fit, unfit, and frail patients at disease onset.
* Malabsorption syndrome or other diseases that affect the ability to swallow oral therapy.
* Concomitant malignancy requiring treatment (except non-melanoma skin cancers and in situ carcinoma of the uterine cervix).
* Presence of opportunistic infections in place.
* Seropositive for or active viral infection with hepatitis B virus (HBV):

  1. HBsAg positive;
  2. HBsAg negative, HBcAb positive with detectable viral DNA (Subjects who are HBsAg negative, HBcAb positive, but viral DNA negative are eligible.
* Seropositive and active infection for hepatitis C virus (subjects who are HCV-RNA negative are eligible).
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV).
* Impossibility to give written informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2020-04-22 (Actual); Study Completion 2021-06-21 (Actual)

PRIMARY OUTCOMES:
Complete Remission Rate (CRR) | 30 months
  The primary efficacy endpoint is defined in terms of complete response (CR), including complete response unconfirmed (CRu), according to Recommendations of an International Workshop to Standardise Response Criteria for Non-Hodgkin´s Lymphomas.
Incidence of adverse events | 30 months
  The primary safety endpoint is defined as incidence, nature, and severity of adverse events graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.03

SECONDARY OUTCOMES:
Overall response rate (ORR) | 30 months
  ORR, defined as the proportion of patients who achieved a CR (including CRu) or a PR.
Clinical Benefit | 30 months
  Defined as the percentage of patients who achieved a CR (including CRu), a PR and a SD.
Progression Free Survival (PFS) | 36
  defined as the time from registration to the first occurrence of progression or relapse or death for any cause other causes than lymphoma, or the date of last follow-up in censored patients.
Event Free Survival (EFS) | 36
  EFS, defined as the time from registration until: early withdrawal, less than CRu, relapse or progression or death by other causes than lymphoma in patients who achieved CR or CRu after the EOI phase.
Disease Free Survival (DFS) | 36
  DFS: calculated for patients in CR/CRu after induction phase, from the date of response/end treatment until relapse, death by other causes than lymphoma or last follow-up in censored patients.
Overall Survival (OS) | 36
  OS, calculated from the date of registration until death for any cause or last follow-up in censored patients.
Patient-Reported Outcome (PRO) | 36
  PRO per European Organization for Research and Treatment of Cancer (EORTC) Quality-of-Life (QLQ-30) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Merli, MD, Principal Investigator — AUSL - IRCCS Arcispedale Santa Maria Nuova viale Risorgimento 80 42123, Reggio Emilia
Locations (10):
- Italy (10):
  - A.O. Spedali Civili di Brescia - Ematologia, Brescia
  - Ospedale di Castelfranco Veneto - Ematologia, Castelfranco Veneto
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.) - Ematologia, Meldola
  - Ospedale Guglielmo da Saliceto - U.O.Ematologia, Piacenza
  - Ospedale delle Croci - Ematologia, Ravenna
  - Azienda Ospedaliera Arcispedale Santa Maria Nuova - IRCCS c/o CORE (II piano) - Ematologia, Reggio Emilia
  - AO Sant'Andrea - Ematologia, Roma
  - Nuovo Ospedale Civile di Sassuolo - Day Hospital Oncologico, Sassuolo
  - AOU Senese - U.O.C. Ematologia, Siena
  - A.O.U. Citta della Salute e della Scienza di Torino - Ematologia Universitaria, Torino

IPD SHARING:
Plan to Share IPD: No